CLINICAL TRIAL: NCT06071156
Title: Serial Cardiac Magnetic Resonance Imaging for Guidance of Therapy Management in Patients Treated With Anakinra Due to Recurrent Pericarditis
Brief Title: Therapy Management in Patients Treated With Anakinra Due to Recurrent Pericarditis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero, Universitaria Ospedali Riuniti (Other)
Responsible Party: Principal Investigator, Francesco Bianco, Cardiologist, Azienda Ospedaliero, Universitaria Ospedali Riuniti
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CCPC- 003/18
Record Dates: First submitted 2023-10-02; First posted 2023-10-06 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Recurrent Pericarditis
Keywords: Anakinra; Cardiac magnetic resonance; Late gadolinium enhancement; C-reactive protein
MeSH Terms: conditions — Pericarditis | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Intervention Model Description: 1:1 randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CMR-guided therapy management, (Active Comparator): The scheme of Anakinra treatment was three months at full dosage, the next three months of therapy at full dosage every other day, and the last three months at halved dosage every other day until the end of treatment. Cardiac magnetic resonance [no pericardial edema and/or late gadolinium enchantment (LGE)] guided each anakinra dose reduction. If the tests were positive for ongoing pericardial inflammation [pericardial edema present or LGE present], the reduction was postponed, and one more month of therapy was administered before the reduction.
  Interventions: Drug: Anakinra
- CRP-guided therapy management, (Active Comparator): The scheme of Anakinra treatment was three months at full dosage, the next three months of therapy at full dosage every other day, and the last three months at halved dosage every other day until the end of treatment. Laboratory tests [C-reactive protein (CRP) <0.6 mg/dL] guided each anakinra dose reduction. If the tests were positive for ongoing systemic inflammation (CRP > 0.6 mg/dL), the reduction was postponed, and one more month of therapy was administered before the reduction.
  Interventions: Drug: Anakinra

INTERVENTIONS:
Drug: Anakinra — Anakinra, an IL-1 antagonist, is particularly interesting because it limits the self-sustained pathway of recurrent pericarditis and may reduce the recurrences

SUMMARY:
To determine the utility of serial cardiac magnetic resonance (CMR) imaging for guidance of therapy management in patients treated with anakinra due to recurrent pericarditis (RP), compared with c-reactive protein (CRP) assay alone.

DETAILED DESCRIPTION:
Recurrent pericarditis (RP) is a specific pathology of the pericardium included within the pericardial syndromes by the guidelines of the European Society of Cardiology (ESC). The latter defines RP as pericarditis occurring after a symptom-free interval of 4-6 weeks from a documented first episode of acute pericarditis; the recurrences rate may range from 15 to 30%, with a significant increment of 50% in patients treated with corticosteroids or not treated with colchicine. The diagnosis of recurrences follows the same criteria utilized for acute pericarditis, and a viral etiology can often be demonstrated.

The pathogenesis of RP is still debated, but they are self-sustained by an autoinflammatory/ autoimmune amplified response following an exogenous or endogenous trigger. In this context, the cytokine interleukin 1 (IL-1) has been implicated as a key mediator of RP. Anakinra, an IL-1 antagonist, is of particular interest because it limits the self-sustained pathway of RP and may reduce the recurrences. The current 2015 ESC guidelines for the diagnosis and management of pericardial diseases recommend anakinra in cases of proven infection-negative, corticosteroid-dependent RP not responsive to colchicine, but it remains debated the duration of the therapy and when to start its tapering. In this context, cardiac magnetic resonance (CMR) imaging has recently emerged as an interesting imaging biomarker capable of detecting pericardial inflammation, proving pericardial edema and late gadolinium enhancement (LGE), and distinguishing three defined pericardial inflammation phases: acute (edema and LGE), subacute (only LGE) and burned-out (no edema nor LGE).

To overcome the 2015 ESC guidelines limitations, the investigators sought to determine the utility of serial CMR imaging for guidance of therapy management in patients treated with anakinra due to RP, compared with the c-reactive protein (CRP) assay alone, as currently recommended.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients treated with anakinra 100 mg/die if ≥ 18 years old, and
* Pediatric patients treated with anakinra 2 mg/kg/die if < 18 years old
* Pediatric and adult patients treated with anakinra due to corticosteroid-dependent or not responsive to colchicine or non-steroidal anti-inflammatory drugs (NSAIDs) recurrent pericarditis

Exclusion Criteria:

* Ongoing infection (proved within serology)
* Refuse to participate in the trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-05-05 (Actual); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Recurrences of pericarditis | 6 month
  Recurrences of pericarditis during Anakinra reduction regimen of therapy

CONTACTS AND LOCATIONS:
Locations (1):
- CCPC, Ancona, The Marches, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Adler Y, Charron P, Imazio M, Badano L, Baron-Esquivias G, Bogaert J, Brucato A, Gueret P, Klingel K, Lionis C, Maisch B, Mayosi B, Pavie A, Ristic AD, Sabate Tenas M, Seferovic P, Swedberg K, Tomkowski W; ESC Scientific Document Group. 2015 ESC Guidelines for the diagnosis and management of pericardial diseases: The Task Force for the Diagnosis and Management of Pericardial Diseases of the European Society of Cardiology (ESC)Endorsed by: The European Association for Cardio-Thoracic Surgery (EACTS). Eur Heart J. 2015 Nov 7;36(42):2921-2964. doi: 10.1093/eurheartj/ehv318. Epub 2015 Aug 29. No abstract available. PMID 26320112
- [Result] Imazio M, Andreis A, De Ferrari GM, Cremer PC, Mardigyan V, Maestroni S, Luis SA, Lopalco G, Emmi G, Lotan D, Marcolongo R, Lazaros G, De Biasio M, Cantarini L, Dagna L, Cercek AC, Pivetta E, Varma B, Berkson L, Tombetti E, Iannone F, Prisco D, Caforio ALP, Vassilopoulos D, Tousoulis D, De Luca G, Giustetto C, Rinaldi M, Oh JK, Klein AL, Brucato A, Adler Y. Anakinra for corticosteroid-dependent and colchicine-resistant pericarditis: The IRAP (International Registry of Anakinra for Pericarditis) study. Eur J Prev Cardiol. 2020 Jun;27(9):956-964. doi: 10.1177/2047487319879534. Epub 2019 Oct 15. PMID 31610707
- [Result] Cremer PC, Lin D, Luis SA, Petersen J, Abbate A, Jellis CL, Kwon D, Brucato A, Fang F, Insalaco A, LeWinter M, Lewis BS, Zou L, Nicholls SJ, Klein AL, Imazio M, Paolini JF; RHAPSODY Investigators. Pericardial late gadolinium enhancement and time to recurrence: a substudy from RHAPSODY, a phase 3 clinical trial of rilonacept in recurrent pericarditis. Eur Heart J Imaging Methods Pract. 2023 May 26;1(1):qyad003. doi: 10.1093/ehjimp/qyad003. eCollection 2023 May. PMID 39044797
- [Result] Conte E, Agalbato C, Melotti E, Marchetti D, Schillaci M, Ratti A, Ippolito S, Pancrazi M, Perone F, Dalla Cia A, Pepi M, Pontone G, Imazio M, Brucato A, Chetrit M, Klein A, Andreini D. The Contemporary Role of Cardiac Computed Tomography and Cardiac Magnetic Resonance Imaging in the Diagnosis and Management of Pericardial Diseases. Can J Cardiol. 2023 Aug;39(8):1111-1120. doi: 10.1016/j.cjca.2023.01.030. Epub 2023 Feb 3. PMID 36740019
- [Result] Kumar A, Sato K, Verma BR, Ala CK, Betancor J, Yzeiraj E, Lin L, Mohananey D, Qamruddin S, Kontzias A, Bolen MA, Imazio MM, Kwon DH, Hachamovitch R, Klein AL. Quantitative assessment of pericardial delayed hyperenhancement helps identify patients with ongoing recurrences of pericarditis. Open Heart. 2018 Dec 16;5(2):e000944. doi: 10.1136/openhrt-2018-000944. eCollection 2018. PMID 30613419
- [Derived] Bianco F, Bucciarelli V, Coretti F, Cataldi S, Damadei F, Raffaelli E, Schicchi N, Omenetti A, Lattanzi B, Berton E, Chiara Surace F, Baldinelli A, Breda L, Cazzato S, Catassi C, Dello Russo A, Gallina S. Serial cardiac magnetic resonance imaging for guidance of therapy management in patients treated with anakinra due to recurrent pericarditis. Eur Heart J Imaging Methods Pract. 2024 Mar 28;2(1):qyae019. doi: 10.1093/ehjimp/qyae019. eCollection 2024 Jan. PMID 39045200